CLINICAL TRIAL: NCT04826549
Title: A Comparison of Exhaled Carbon Monoxide Measurements Using the iCOquit Smokerlyzer and Vitalograph Breath CO Monitor vs Carboxyhemoglobin From Venous Samples While Validating a Mobile Research Application
Acronym: COCO
Status: Completed | Type: Observational
Sponsor: Rose Research Center, LLC (Industry)
Collaborators: Foundation for a Smoke Free World INC (Other)
Responsible Party: Sponsor
Other Study IDs: COCO
Record Dates: First submitted 2021-03-26; First posted 2021-04-01 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Smoking, Cigarette
MeSH Terms: conditions — Cigarette Smoking

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of this study is to determine the accuracy and precision of the iCOquit Smokerlyzer as compared with the gold standard of COHb levels measured in venous plasma samples, as well as assessing its agreement with the Vitalograph BreathCO monitor. Validating the precision and accuracy of the iCOquit Smokerlyzer could establish an additional, less expensive, reliable method for determining smoking status in tobacco research. Additionally, the portability of the device would allow for remote biochemical verification of smoking status, thus enlarging the number of participants that can be included in intervention studies.

ELIGIBILITY:
Inclusion Criteria:

1. Has signed the ICF and is able to read and understand the information provided in the ICF.
2. Is 21 to 65 years of age (inclusive) at screening.
3. No intention of quitting smoking in the next 30 days.
4. Willing and able to comply with the requirements of the study.
5. Owns a smartphone running iOS or Android with text message and data capabilities compatible with the eResearch app.

Exclusion Criteria:

1. Is unhealthy or cannot participate in the study for any reason (e.g., medical, psychiatric, and/or social reason) as judged by the Investigators or designated medical staff based on all available assessments from the screening period (e.g., vital signs, physical examination, concomitant medications and medical history).
2. PHQ-9 score greater than 9, or a score greater than 0 on item #9 ("Thoughts you would be better off dead, or of hurting yourself in some way") at screening.
3. Body mass index (BMI) greater than 40.0 kg/m2
4. Use of any of these products in the past 30 days:

   1. Illegal drugs (or if the urine drug screen is positive for cocaine, THC, amphetamines, methamphetamines, or opiates),
   2. Experimental (investigational) drugs that are unknown to participant,
   3. Chronic opioid use.
5. Pregnant or nursing (by self-report) or positive urine pregnancy test.
6. Participant enrollment numbers met.

   -

Ages: 21 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Combustible cigarette smokers from Raleigh, NC and Charlotte, NC and surrounding areas.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2021-10-27 (Actual)

PRIMARY OUTCOMES:
eCO Monitor Accuracy compared to COHb | Baseline
  Determine the accuracy and precision of the iCOquit Smokerlyzer as compared with the gold standard of COHb levels measured in venous plasma samples.
eCO Monitor's agreement with the Vitalograph BreathCO monitor | Baseline
  Comparing the CO values from the eCO Monitor and the Vitalograph BreathCO monitor.

SECONDARY OUTCOMES:
eRESEARCH APP VALIDATION | Daily for 5 days
  Validate a new mobile app called eResearch through specific functionality testing by study participants.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Rose Research Center, Charlotte, North Carolina
  - Rose Research Center, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: No